CLINICAL TRIAL: NCT00926198
Title: Frequency, Pathogen Spectrum and Specific Immune Response in Acute Pharyngotonsillitis in Children and Adolescents
Brief Title: Investigation of Clinical Spectrum, Bacterial Pathogens and Immune Response in Acute Pharyngotonsillitis
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Prof. Stefan Zielen, Medaimun GmbH and Johann Wolfgang Goethe University Hospitals
Other Study IDs: KGU- 31/09
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Tonsillitis
Keywords: Upper airway infections; pharyngotonsillitis; GABHS
MeSH Terms: conditions — Tonsillitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — throat culture, blood sample
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute pharyngotonsillitis is one of the most common infections encountered by pediatricians. Most children with acute pharyngotonsillitis have symptoms that can be attributed to viral infection. However 30-40% of cases is of bacterial etiology.

The purpose of this study is to examine frequency, age distribution, clinical picture and pathogen distribution in acute pharyngotonsillitis in children in a large urban setting.

DETAILED DESCRIPTION:
According to the US Vital Health Statistics report, acute pharyngotonsillitis is responsible for more than 6 million office visits each year by children younger than 15 years of age. Approximately 30% of cases is of bacterial etiology and group A beta-hemolytic streptococci(GABHS) are responsible for most bacterial cases, although other pathogens, such as Neisseria gonorrhoeae, Arcanobacterium haemolyticum, Mycoplasma pneumoniae, and Chlamydia pneumoniae, may be the causative agents in sporadic cases. An accurate diagnosis of GABHS infection is important because it is the only common form of acute pharyngotonsillitis for which antibiotic therapy is definitely indicated. Effective antibacterial treatment can shorten the clinical course of GABHS pharyngotonsillitis, reduce the rate of transmission, and prevent suppurative and nonsuppurative complications, such as peritonsillar abscess and acute rheumatic fever.

This study enrolls patients who will present with acute fever and clinical signs of pharyngotonsillitis at three primary pediatric ambulances. A rapid A beta-hemolytic streptococcus (GABHS)-detection test will be performed in these patients. In one office, additional throat cultures are obtained of all patients, and blood is taken in a subgroup of 60 GABHS-positive and 60 GABHS-negative cases. In GABHS-positive patients, a second blood sample will be obtained at day 7th and day 28th, and stored until specific antibody response to GABHS will be measured.

ELIGIBILITY:
Inclusion Criteria:

* age 3 months to 18 years
* clinical signs of tonsillopharyngitis
* informed consent

Exclusion Criteria:

* age more than 18 years
* diagnosed chronic disease or infection (e.x. HIV, tuberculosis, malignancy)
* current participation in another research projects that may interfere with this study
* Incapability to perform all study procedure

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 3 months to 18 years who will present clinical signs of tonsillopharyngitis.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The responsible pathogens (Frequency of GABHS) of acute pharyngotonsillitis and its clinical and serological response in children in a large urban setting. | 1 year

SECONDARY OUTCOMES:
In a subset of patients the immune response to GABHS will be measured at beginning and after 7 and 28 days. | one month

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Prof., Principal Investigator — Medaimun GmbH and Johann Wolfgang Goethe University
Locations (3):
- Germany (3):
  - Paeditric office, Babenhausen, Hesse
  - Paediatric office, Dietzenbach, Hesse
  - Paediatric office, Offenbach-Rumpenheim, Hesse

REFERENCES:
- [Background] Shulman ST. Acute streptococcal pharyngitis in pediatric medicine: current issues in diagnosis and management. Paediatr Drugs. 2003;5 Suppl 1:13-23. PMID 14632102
- [Background] Brook I, Dohar JE. Management of group A beta-hemolytic streptococcal pharyngotonsillitis in children. J Fam Pract. 2006 Dec;55(12):S1-11; quiz S12. PMID 17137534
- [Background] Nussinovitch M, Finkelstein Y, Amir J, Varsano I. Group A beta-hemolytic streptococcal pharyngitis in preschool children aged 3 months to 5 years. Clin Pediatr (Phila). 1999 Jun;38(6):357-60. doi: 10.1177/000992289903800606. PMID 10378093